CLINICAL TRIAL: NCT06695078
Title: Nutrition in Paediatric Critical Care: a Bi-national Prospective Cohort Study
Brief Title: Nutrition in Paediatric Critical Care
Acronym: ePICUre
Status: Recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/JW001
Record Dates: First submitted 2024-10-28; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: ICU; Nutrition; Paediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
This is a multi-centre prospective cohort study of nutrition in paediatric critical care in Australia and New Zealand. The study is planned to run in parallel with the adult ICU cohort study, NUTRIENT. Two study periods are proposed with the first in late 2024 and the second in 2026. This observational study seeks to determine the following (although not limited to) descriptive outcomes of interest:

1. Nutritional outcomes, including route of nutrition support (oral, enteral and/or parenteral), energy and protein prescription and provision, and anthropometric measures
2. Patient-centred outcomes, including duration of invasive respiratory support and hospitalisation, and mortality
3. Nutrition service delivery in the PICU and ward settings

ELIGIBILITY:
Inclusion Criteria:

1. All patients </=18 years of age
2. Admitted to the PICU after 00:00 on the day of the study period commencement
3. Admitted to the PICU for >72 hours

Exclusion Criteria:

1. Those previously enrolled during the study period (i.e. those re-admitted to PICU)
2. Those for end of life care only
3. Those admitted for organ donation

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children aged under 18 years admitted for >72 hours to participating PICUs during the two-week study recruitment period. Further funding will be sought to continue this study beyond the 2026 data collection period.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-07 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Energy intake as proportion of estimated requirements | Up to day 28 of hospitalization
  Oral, enteral and parenteral energy intake will be collected and reported as a proportion of estimated requirements; estimation of requirements will be standardised using the Schofield equation and dependent upon the reported phase of critical illness

SECONDARY OUTCOMES:
Protein intake as proportion of estimated requirements | Up to day 28 of hospitalization
  Oral, enteral and parenteral protein intake will be collected and reported as a proportion of estimated requirements; estimated requirements will be standardised and dependent upon reported phase of critical illness
Route of nutrition provision | Up to day 28 of hospitalization
  Data will be collected on route of nutrition provision (oral, enteral or parenteral); enteral route will be categorised according to type of enteral feeding route
Type of nutrition provision (type of diet or oral/enteral feed/formula) | Up to day 28 of hospitalization
  Data will be collected on the type of nutrition provision, in regards to type of diet and the type of formula or feed provided orally or enterally
Anthropometric measures reported as z-scores | Up to day 28 of hospitalization
  Weight and length/height will be collected (and head circumference for children up to 2 years gestational age); these measures will be reported according to WHO growth standard z-score (up to 2 years age) or CDC growth standard z-scores (2 years age and above)
Multidisciplinary nutrition assessment and intervention | Up to day 28 of hospitalization
  Data will be collected on the frequency of nutrition assessment or intervention, including which profession completed the assessment or intervention (i.e. dietetics, medical, nursing or other)
Duration of invasive ventilation | Up to day 28 of hospitalization
  Data will be collected on the duration of invasive ventilation
Duration of PICU and hospital admission | Up to day 28 of hospitalization
  Duration of PICU and overall hospital admission will be collected

CONTACTS AND LOCATIONS:
Locations (11):
- Australia (10):
  - Women's and Children's Hospital Adelaide, Adelaide
  - Queensland Children's Hospital, Brisbane
  - Royal Hobart Hospital, Hobart
  - Monash Children's Hospital, Melbourne
  - The Royal Children's Hospital Melbourne, Melbourne
  - Perth Children's Hospital, Perth
  - Sunshine Coast Hospital, Sunshine Coast
  - John Hunter Children's Hospital, Sydney
  - Sydney Children's Hopsital, Sydney
  - The Children's Hospital at Westmead, Sydney
- Starship Children's Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No